CLINICAL TRIAL: NCT04939935
Title: Implementation of Metformin theraPy to Ease Decline of Kidney Function in Polycystic Kidney Disease (IMPEDE-PKD): A Randomised Placebo-Controlled Trial
Brief Title: Implementation of Metformin theraPy to Ease Decline of Kidney Function in Polycystic Kidney Disease (IMPEDE-PKD)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKTN16.01
Record Dates: First submitted 2021-06-16; First posted 2021-06-25 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-07

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Placebo; Metformin; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomised to either (1) intervention group receiving metformin extended release (XR) plus standard of care, or (2) placebo plus standard of care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study participants, treating physicians and other care providers, outcome assessors, study investigators, and study statisticians will be blinded. An unblinded statistician will regularly review treatment allocations to ensure balance across treatment arms. The unblinded statistician will also prepare unblinded statistical reports for meetings of the Data and Safety Monitoring Board.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants randomised to the intervention group receive Metformin XR plus standard of care for 104 weeks.
  Dosage will depend on individual participant's level of tolerance to Metformin XR as well as their estimated glomerular filtration rate (eGFR). The dosage will be between 500-2000mg/day.
  Interventions: Drug: Metformin XR
- Control (Placebo Comparator): Participants randomised to the control group receive placebo plus standard of care for 104 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Metformin XR — Extended release metformin.
  Other Names: APO-Metformin XR (500mg)
  Arms: Intervention
Other: Control — Placebo is inactive tablets that is identical to the intervention Metformin tablets.
  Other Names: Placebo
  Arms: Control

SUMMARY:
This study will investigate if a medication (metformin) widely used in the treatment of diabetes could be re-purposed for the treatment of patients with a diagnosis of early stage ADPKD to slow the rate of kidney function decline, reducing morbidity and mortality and improving the quality of life for ADPKD patients.

DETAILED DESCRIPTION:
Autosomal Dominant Polycystic Kidney Disease (ADPKD) affects 12.5 million people worldwide and is the 4th leading cause of kidney failure. Cyst growth begins in childhood, and over decades leads to painful kidneys, hypertension and chronic kidney disease. ADPKD patients also have a high prevalence of anxiety, depression and poor quality of life. Despite this enormous burden, there is a lack of evidence for therapies and affordable, effective treatment options. To date, only one disease modifying therapy is licensed for use in ADPKD (tolvaptan), but it is limited by its restricted availability, side effects and high cost. Metformin, an inexpensive and familiar drug, has been shown in previous studies to target cyst-forming signals, thereby slowing the cyst growth rate. IMPEDE-PKD is an Australian-led global Phase III randomised controlled trial to investigate the effect of metformin on ADPKD disease progression. The study will recruit a total of 1,174 adult ADPKD patients from around the world (250 from Australia). The outcomes of this research will identify effective and targeted therapies for ADPKD that will slow kidney function decline, reduce the impact of the illness and likelihood of death, and improve the quality of life for ADPKD patients and families.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, patients must satisfy all of the following inclusion criteria:

1. Willing to participate and provide informed consent
2. Aged 18-70 years
3. Diagnosis of ADPKD based on radiological +/- genetic criteria as per Kidney Health Australia - Caring for Australians and New Zealanders with Kidney Impairment (KHA-CARI) Guidelines
4. eGFR equal to or greater than 38 mL/min/1.73m2 and <90 mL/min/1.73m2

And have either:

5(a) One or more risk factors of progression from the following:

* Bilateral kidney length equal to or greater than16.5 cm, or
* Total Kidney Volume (TKV) equal to or greater than 750 mL or height-adjusted TKV (htTKV) equal to or greater than 600 mL/m2, or
* Mayo class IC/D/E or Pro-PKD score equal to or greater than 6 OR 5(b) Evidence of Active progression
* Decline in eGFR equal to or greater than 5 mL/min/1.73m2 in one year, or
* Decline in eGFR equal to or greater than 3 mL/min/1.73m2 per year over five years or more. or
* Increase in htTKV/TKV of equal to or greater than 5% per year on at least 2 measurements in the past year, excluding any initial eGFR effect over the initial 3 months of tolvaptan commencement (if applicable) Note: Tolvaptan therapy must have been in place for at least 6 months with stable dose for at least 3 months.

Exclusion Criteria:

1. Diabetes mellitus (as per American Diabetes Association definition), or other systemic conditions that may cause CKD independent of PKD (excluding hypertension)
2. Uncontrolled hypertension (Systolic BP >160 mmHg and/or diastolic BP >100 mmHg after a period of rest)
3. Clinically significant heart failure, including but not limited to New York Heart Association Class (NYHA) III or IV
4. Non-polycystic liver disease, including but not limited to:

   1. Liver enzymes (ALT, AST or Total Bilirubin) >2 times the upper limit of normal, except when a diagnosis of Gilbert Syndrome exists and/or,
   2. Child-Pugh classification score equal to or greater than 5
5. Any contraindication to metformin including abnormal liver function tests or untreated Vitamin B12 deficiency
6. Currently taking metformin
7. Pregnancy or breastfeeding, or planning to get pregnant in the next three years.
8. Comorbidities with potential to contaminate trial outcomes, specifically active cancer, history of other solid organ transplantations, active chronic obstructive pulmonary disease (COPD), active inflammatory bowel disease, and the presence of stoma.
9. History of dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1174 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The change in estimated glomerular filtration rate (eGFR) | Over 24 months
  This will be measured using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula at 104 weeks (24 months) from first dispensing date.

SECONDARY OUTCOMES:
Annualised slope of eGFR. | Over 24 months
  The mean rate of change in eGFR from baseline over 2 years, estimated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula from the serum creatinine concentration analysed in the central laboratory.
Composite outcome | Over 24 months
  A composite outcome comprising a reduction from baseline eGFR of equal to or greater than 30%, kidney failure (defined as an eGFR <15 millilitres/min/1.73m2), and all-cause mortality.
Severity of change in eGFR | Over 24 months
  The proportion of participants with a reduction from baseline in their eGFR of equal to or greater than 30%.
Kidney failure | Over 24 months
  The proportion of participants who experience kidney failure, defined as an eGFR <15mL/min/1.73m2.
Mortality | Over 24 months
  The proportion of participants who die during the observation period, irrespective of the cause.
Change in medication dosage during the trial | Over 24 months
  The proportion of participants requiring a dosage increase or the introduction of a new anti-hypertensive agent during the treatment period.
Changes in the urine albumin:creatinine ratio | Over 24 months
  The percentage change in the urine albumin:creatinine ratio for each participant
Presence and category change of albuminuria | Over 24 months
  The proportion of participants who experience albuminuria (excess albumin in the urine) during the trial period. Raw values will be recorded and albuminuria will be categorised as either A1 (<3.39mg/mmol), A2 (3.39-33.9mg/mmol), or A3 >33.9mh/mmol.
Health-related quality of life | Over 24 months
  This will measured using the EuroQual 5 Domain 5 Level (EQ-5D-5L) questionnaire
ADPKD-related pain | Over 24 months
  Mean change in the ADPKD Pain and Discomfort Scale (ADPKD-PDS) from baseline to end of study (dull kidney pain, sharp kidney pain and fullness/discomfort domain scores will be reported and analysed).
Gastrointestinal symptoms | Over 24 months
  This will be measured using the Gastrointestinal Symptom Rating Scale (GSRS). A score greater than 1.33 will signal the presence of patient-significant gastrointestinal symptomatology
Presence of study-related events | Over 24 months
  The proportion of participants who experience a specific event related to the study treatment (sub-categorised as incidence of gastrointestinal symptoms, presence of lactic acidosis, deranged liver function tests, hypoglycaemia, anaemia and vitamin B12 deficiency) expressed as a rate per 100 person years
Healthcare utilisation | Over 24 months
  Incremental cost effectiveness ratios (ICERs) will be calculated based on the incremental costs and incremental health outcomes between intervention groups

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Mallett, MBBS, PhD, Principal Investigator — Townsville University Hospital
Locations (40):
- Australia (13):
  - Renal Research, Gosford, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital - Western Sydney Local Health District, Sydney, New South Wales
  - Bundaberg Hospital, Bundaberg, Queensland
  - Townsville University Hospital, Douglas, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- New Zealand (4):
  - Te Whatu Ora - Hauora a Toi Bay of Plenty, Tauranga, Bay of Plenty
  - Te Whatu Ora - Te Tai Tokerau, Whangārei, Northland
  - Te Whatu Ora - Southern, Dunedin, Otago
  - Te Whatu Ora - Taranaki, New Plymouth, Taranaki Region
- United Kingdom (23):
  - Royal Devon & Exeter Hospital, Exeter, Devon
  - Nottingham Renal Unit, Nottingham City Hospital, Nottingham, East Midlands
  - Raigmore Hospital, Inverness, Inverness Shire
  - Royal Preston Hospital, Preston, Lancashire
  - Salford Royal Hospital, Salford, Lancashire
  - Leicester General Hospital, Leicester, Leicestershire
  - St Helier Hospital, Carshalton, London
  - The Royal London Hospital, London, London
  - Royal Free Hospital, London, London
  - King's College Hospital, London, London
  - Aintree University Hospital, Liverpool, Merseyside
  - Norfolk and Norwich University Hospital, Norwich, Norfolk
  - Antrim Area Hospital, Antrim, Northern Ireland
  - Ulster Hospital, Belfast, Northern Ireland
  - Altnagelvin Hospital, Londonderry, Northern Ireland
  - Daisy Hill Hospital, Newry, Northern Ireland
  - Oxford Kidney Unit, Churchill Hospital,, Oxford, Oxfordshire
  - Doncaster Royal Infirmary, Doncaster, South Yorkshire
  - Sheffield Kidney Institute, Sheffield, South Yorkshire
  - Royal Stoke University Hospital, Stoke-on-Trent, Staffordshire
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear
  - Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands
  - Bradford Renal Unit, St Luke's Hospital, Bradford, West Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cortinovis M, Perico N, Remuzzi G. The Need for Novel Therapeutic Directions in Autosomal Dominant Polycystic Kidney Disease Patient Care. Clin J Am Soc Nephrol. 2025 Dec 5. doi: 10.2215/CJN.0000000975. Online ahead of print. PMID 41348481
- [Derived] Pierre KS, El-Damanawi R, Johnson DW, Hawley CM, Viecelli AK, Jha V, Green SC, Gesualdo L, Kiriwandeniya C, Velayudham P, Vergara LA, Mihala G, Matsuyama M, Brent PP, Mallett AJ; IMPEDE-PKD Global Steering Committee (see Appendix). Implementation of Metformin Therapy to Ease Decline of Kidney Function in Polycystic Kidney Disease (IMPEDE-PKD): study protocol for a phase III, multi-centre, randomized, placebo-controlled trial evaluating the long-term efficacy of metformin in slowing the rate of kidney function decline in patients with autosomal dominant polycystic kidney disease. Trials. 2025 Aug 25;26(1):302. doi: 10.1186/s13063-025-09010-6. PMID 40855441
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] El-Damanawi R, Stanley IK, Staatz C, Pascoe EM, Craig JC, Johnson DW, Mallett AJ, Hawley CM, Milanzi E, Hiemstra TF, Viecelli AK. Metformin for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2024 Jun 4;6(6):CD013414. doi: 10.1002/14651858.CD013414.pub2. PMID 38837240